# Influence of Financial Incentives on Oral Disease Management in Young Children (BEhavioral EConomics for Oral health iNnovation - BEECON)

**NIDCR Protocol Number: 17-084-E** 

**NIDCR Grant Number: UH3DE025514** 

ClinicalTrials.Gov Number: NCT03576326

UCSF IRB Number: 17-23786

ICF Version Number: 1.3

ICF Date: 15 August 2018

ICF Language: Spanish

# CONSENT FOR PARENT AND PARENTAL PERMISSION FOR MINOR TO PARTICIPATE IN RESEARCH STUDY (SPANISH)

University of California, Los Angeles (UCLA) and the University of California, San Francisco

BEECON TRIAL - Influence of Financial Incentives on Oral Disease Management in Young Children (BEhavioral EConomics for Oral health iNnovation)

# ¿Qué es los que deseamos aprender del estudio?

Un equipo de dentistas y científicos desean estudiar 1) las actitudes de los padres sobre la salud oral de sus hijos y 2) ayudar a los padres a detener las caries en niños pequeños, al cepillar los dientes de los niños y llevar a los niños al dentista.

Para participar en este estudio,

## Su hijo/a debe tener:

- · Al menos 6 meses, pero menos de 4 años;
- Con al menos dos dientes completamente en su boca;
- Inscrito o en lista de espera para uno de los programas participantes de Early Head Start de Los Ángeles o un programa de guardería afiliado;
- Libre de alergias a los productos del estudio, incluyendo el líquido de revelación de placas o el barniz de fluoruro;
- Capaz de abrir su boca sin ayuda para permitir que el dentista mire sus dientes, los limpie y permita que los asistentes de investigación fotografíen los dientes.
- Sin más de 2 coronas en los dientes de los incisivos maxilares (#D, E, F, G, o equivalente #52, 51, 61, 62).

#### Usted, el padre o guardián, debe:

- Ser el cuidador principal del niño que cepillará los dientes del niño todos los días (desafortunadamente, los niños de crianza temporal no son elegibles);
- Planee vivir en el área de Los Ángeles durante los próximos 18 meses:
- Tener un "Smart Phone" y estar dispuesto a descargar y mantener una aplicación gratuita desde Google Play o Apple Store durante la duración del proyecto; y,
- Estar dispuesto a que el personal del estudio se comunique con usted por SMS (mensajes de texto) para mandarle mensajes sobre el estudio.

Habrá 240 niños con sus padres en este estudio. Los padres serán colocados en uno de los dos grupos al azar por computadora (como lanzar una moneda o lanzar un dado) que tendrá las mismas oportunidades, pero en diferentes momentos durante el programa.

Este estudio está siendo pagado por los Institutos Nacionales de Salud.

# ¿Qué sucederá si tomamos parte en este estudio de investigación?

Este estudio durará hasta 18 meses. Si usted y su hijo se ofrecen como voluntarios para unirse a este estudio, le pediremos que haga lo siguiente:

# EN LA PRIMERA VISITA DEL ESTUDIO (PRIMER ESTUDIO) (60-90 min):

- Se le harán preguntas sobre la salud oral de su hijo, las visitas dentales anteriores y las actitudes, comportamientos y conocimientos dentales de su familia. Mantendremos sus respuestas y archivos confidenciales en una computadora. El equipo combinará estas respuestas con otras familias
- Se le pedirá que vea un video sobre la salud oral.

- Su hijo tendrá un examen dental y un líquido de revelación rojo pintado en los dientes de su hijo para verificar su nivel de placa. Se tomará una fotografía de los dientes y se conservará en el archivo de estudio dental de su hijo. Las fotos podrán ser usadas para presentaciones, publicaciones o propósitos de investigación, pero no identificarán a su hijo ni publicarán el nombre de usted ni el de su hijo.
- Además, el barniz de fluoruro se pintará en los dientes de su hijo para protegerlos de las caries dentales.
- Aprenderá a cepillar los dientes de su hijo con un cepillo especial de dientes eléctrico le daremos a su hijo. Con nuestra ayuda, instalará una aplicación gratuita en su "Smart Phone", que se conectara con el cepillo de dientes del estudio y observará qué tan bien le está lavando los dientes a su hijo.

# EN CASA, se le pedirá que:

- Practique cepillando los dientes de su hijo cada mañana y cada noche durante 1 minuto cada vez con el cepillo de dientes eléctrico y la pasta de dientes que le darán en la primera visita.
- Sincronice el cepillo de dientes eléctrico con la aplicación de su teléfono tres veces a la semana durante 2 semanas. Se le pagará \$1 por sincronizar el miércoles, viernes y domingo hasta \$3 por semana.

# EN LA SEGUNDA VISITA DEL ESTUDIO (Aproximadamente dos semanas después, 60 minutos):

- Veremos cómo le fue en casa con la aplicación en su "Smart Phone" y el cepillado con el cepillo especial. Si desea continuar, será colocado en uno de los dos grupos al azar por una computadora. Esto significa que ni usted ni nuestro personal pueden elegir el grupo para usted y su hijo.
  - Grupo 1: Sera entrado a un sorteo semanal para cepillar los dientes de los niños regularmente durante seis meses. Luego, seguirá cepillando los dientes de su hijo regularmente durante seis meses adicionales sin recompensas por un tiempo total de proyecto de 12 meses.
  - Grupo 2: No será elegible para premios o sorteos durante los primeros 12 meses, pero podrá ganar recompensas de dibujo más tarde durante los meses 13-18 por usar el cepillo con regularidad.

## EN CASA, se le pedirá que:

- Cepille los dientes de su hijo cada mañana y cada noche durante 1 minuto cada vez con el cepillo de dientes eléctrico y la pasta de dientes que le darán en la primera visita.
- Sincronice el cepillo de dientes eléctrico con la aplicación de su teléfono tres veces por semana durante 3 meses. Se le pagará \$1 por sincronizar en cada uno de estos días: miércoles, viernes y domingo hasta \$3 por semana.

#### **VISITAS FUTURAS**

Después de las dos primeras visitas de estudio, usted y su hijo participarán en este estudio durante aproximadamente 12-18 meses (1-1.5 años) según el grupo al que se le haya asignado alzar.

Habrá al menos 6 visitas en total, incluyendo su primera visita. Nos veremos cada 3 meses y veremos a su hijo dos veces al año para revisiones dentales (aproximadamente cada 6 meses). Después de 12 semanas (3 meses), nos veremos para su primera cita de seguimiento.

- Las visitas de 3 meses, 9 meses y 15 meses (si corresponde) durarán aproximadamente 45 minutos.
- Las visitas de 6 meses, 12 meses y 18 meses (si corresponde) durarán aproximadamente 60 minutos, incluyendo una evaluación dental y una aplicación de barniz de fluoruro para su hijo.

- Se le harán preguntas similares sobre la salud oral de su hijo, las visitas dentales y las actitudes, comportamientos y conocimientos dentales de su familia.
- Se le pedirá que vea un video sobre la salud oral.
- En las visitas de evaluación dental, se pintará un líquido rojo en los dientes de su hijo para notar su nivel de placa. Se tomará una fotografía de los dientes y se conservará en el archivo del estudio dental de su hijo/a.
- En las visitas de seguimiento, recibirá cabezales de cepillo dental adicionales, pasta de dientes (cada 6 meses), sincronización y pagos de visita y recompensas obtenidas (si corresponde).

# INFORMACIÓN IMPORTANTE SOBRE TODAS LAS VISITAS DEL ESTUDIO:

- No tomaremos radiografías. Si el dentista del estudio piensa que su hijo necesita tratamiento dental, recomendaremos que lleve a su niño/a a una clínica dental o a su dentista regular para su evaluación y tratamiento.
- Es posible que su hijo no vea al mismo dentista o asistente dental en cada visita.

Si está inscrito en Early Head Start, la fecha de sus visitas dentales recientes de su hijo se obtendrán del programa de mantenimiento de registros de Early Head Start.

# ¿Cuánto tiempo tomará este estudio de investigación?

El estudio incluirá 6-8 visitas de estudio en persona. En casa, solo le tomará unos minutos para sincronizar el cepillo de dientes eléctrico con su aplicación de "Smart Phone" y solo tomará unos minutos a la semana leer mensajes de texto SMS del estudio.

Si está inscrito en el Grupo 2, tendrá la oportunidad de obtener recompensas después de los 12 meses iniciales y recibirá sus recompensas en las visitas de seguimiento de 15 meses y 18 meses. Si está en el Grupo 2 y decide continuar, será colocado de nuevo en uno de los dos grupos al azar por computadora (como lanzar una moneda o lanzar un dado) que tendrá el mismo número de oportunidades para recibir las mismas recompensas; un grupo será elegible para los sorteos semanales y se les contará semanalmente; el otro grupo será elegible para 13 sorteos cada 3 meses y se lo contará cada 3 meses.

Podrá ser invitado a una discusión de grupo de enfoque que ocurrirá en español o inglés, y puede elegir el idioma que prefiera. Durante la discusión grupal, el facilitador presentará algunos temas y permitirá que los padres hablen libremente sobre sus opiniones y sugerencias. La discusión de grupo será grabada en audio para que el equipo de investigación luego pueda revisar cuidadosamente lo que se ha dicho. La discusión del grupo de enfoque durará aproximadamente 2 horas.

Como esta es una discusión en grupo, otros en el grupo sabrán lo que dirás Mantendremos confidencial la información que nos diga, y no la compartiremos de manera que se pueda identificar.

Participación en el estudio es voluntario. No afectará su relación futura o actual con la Venice Family Clinic Westside Children's Center, Early Head Start, Mujeres, Bebés y Niños, la Universidad de California en San Francisco, la Universidad de California en Los Ángeles o el cuidado médico o dental de su hijo. Puede dejar de participar en cualquier momento sin penalización; no perderá ninguna guardería ni beneficios de salud para usted o su hijo si decide retirarse.

¿Existen posibles riesgos o incomodidades que podamos esperar de este estudio? La solución de revelación de la placa roja (marca GUM Red-Cote Liquid), el barniz de fluoruro (3M ESPE Vanish) y la pasta de dientes con fluoruro (marca Colgate) no han mostrado ningún riesgo o incomodidad con el uso de estos productos dentales. En el raro caso de una reacción alérgica, es posible que su hijo sufra una breve inflamación de las encías, problemas para respirar en niños con asma o náuseas o vómitos en algunos niños que toman demasiado fluoruro. En la rara ocasión de que esto ocurra, se le recomienda llevar a su hijo a un médico para que lo atiendan. Si su hijo ha tenido este tipo de reacción al barniz de fluoruro en el pasado, no puede participar en este estudio. El líquido revelador de placa roja y el barniz de fluoruro será pintado en los dientes de su hijo. Si no es usado de acuerdo a las instrucciones, el cepillo electrónico podría causar molestias en las encías o dientes de su hijo/a. En casos raros, las cerdas de los cabezales del cepillo podrán caerse y ser un obstáculo; dígale a su hijo que no mastique la cabeza del cepillo.

Mantenga la pasta de dientes con flúor fuera del alcance de los niños pequeños para que solo se use la dosis correcta (unte un poco para niños menores de 3 años o tamaño de guisantes para niños de 3 años en adelante).

*Riesgos desconocidos*: los investigadores le informarán si aprenden algo sobre estos productos que podrían hacerle cambiar de opinión acerca de su participación en el estudio.

Algunas preguntas en la encuesta pueden hacer que se sienta incómodo. Puede optar por no responder a ninguna pregunta que no desee responder.

## ¿Hay algún beneficio potencial si participamos?

Los beneficios incluyen una evaluación dental, aplicación de barniz de fluoruro, educación de la salud oral y herramientas del cepillado dental, como cepillo de dientes eléctrico y pasta de dientes. La información que nos dé nos ayudará a comprender maneras de mejorar la atención de la salud oral para los niños pequeños y ayudar a su hijo a tener una mejor salud dental y menos caries.

Su hijo recibirá el chequeo dental y la aplicación de barniz de fluoruro del proveedor dental sin costo para usted.

# ¿Se nos pagará por participar?

Por su tiempo, esfuerzo y gastos de viaje, recibirá un cupón de regalo para el supermercado de \$30 por cada visita de estudio completada.

# ¿Se mantendrá confidencial la información sobre nuestra participación?

Se harán todos los esfuerzos posibles para mantener su información personal privada y confidencial. El equipo de investigación tendrá acceso a la información sobre usted y su hijo, pero los nombres, direcciones, números de teléfono e información de fecha específica no se usarán en ningún informe. Sin embargo, si usted o un miembro de su familia cambia el perfil de la aplicación del número de identificación del estudio al nombre del niño/a, estos datos serán enviados a Philips/Sonicare.

Las organizaciones autorizadas pueden observar los hábitos de cepillado seguidos por el cepillo de dientes eléctrico para la investigación, la precisión y el análisis de datos; estos incluyen Philips Oral Healthcare, y las Juntas de Revisión Institucional de UCSF y UCLA. Otras agencias gubernamentales involucradas en mantener la investigación a salvo para personas como el Instituto Nacional de Investigación Dental y Craneofacial (NIDCR, por sus siglas en inglés), un componente de los Institutos Nacionales de Salud (NIH) y la Administración de Drogas y Alimentos (FDA) pueden ver los datos. Otro personal de la Universidad de California también podrá necesitar que revisar los registros de, o recibir información sobre, participantes

individuales y podrán ver el nombre de usted o el de su hijo. Todos los que tengan acceso a sus archivos mantendrán la información confidencialmente como lo permita la ley.

Acceso a los registros del estudio: La información individual de la evaluación dental de su hijo solo estará disponible para el médico o el dentista en caso de un problema de salud para darle la mejor atención médica a su hijo. Cuando termine el estudio, podrá obtener una copia de los resultados del estudio, pero no los datos o registros individuales de su hijo.

Mantención de registros del estudio: El Dr. Ramos-Gomez, el Dr. Gansky y su equipo de investigación mantendrán sus registros en su oficina. Los registros de menores serán retenidos de acuerdo con las recomendaciones del NIH, o si no se establece ninguna guía, de acuerdo con la recomendación del Consejero General de la UC, que es que los registros se conserven durante 7 años después de que un niño cumpla 18 años (la mayoría de edad), o hasta que el niño tenga 25 años. Esto podría significar que los registros de su hijo se mantendrían en formato digital hasta 25 años después del final del estudio. La información de salud personal de su hijo no puede usarse para investigaciones adicionales sin la aprobación adicional de usted o un comité de revisión.

# ¿Cuáles son los costos de participar en este estudio?

Para enviar notificaciones y recordatorios, a menos que su plan telefónico tenga textos ilimitados, se pueden aplicar tarifas estándar de mensajes de texto SMS.

# ¿A quién puedo contactar si tengo preguntas sobre este estudio?

# El equipo de investigación:

La persona que firme a continuación, y que le explicó el estudio, puede responder cualquier otra pregunta. La línea telefónica del proyecto es (424) 371-6725 y el asistente de investigación puede responder cualquier pregunta en español o inglés. También puede llamar a la gerente de proyectos del estudio, Helen Lindau, al (310) 825-3477. También puede comunicarse con el Dr. Francisco Ramos-Gomez, que es bilingüe en español e inglés, al (310) 825-9460 en Los Ángeles, o al Dr. Stuart Gansky al (415) 502-8094 en San Francisco.

Si tiene preguntas sobre sus derechos como sujeto humano y participante en este estudio, puede llamar a la oficina del Consejo de Revisión Institucional de la Universidad de California, San Francisco al (415) 476-1814.

#### CONSENTIMIENTO

Las Juntas Institucionales de Revisión de UCSF y UCLA han aprobado este formulario de consentimiento, que se indica mediante el sello de las Juntas. Puede solicitar ver los sellos de aprobación de las Juntas en cualquier momento de cualquier miembro del equipo de estudio. El formulario de consentimiento debe revisarse anualmente y expira en la fecha indicada en el sello.

Si su hijo se lesiona como resultado de estar en este estudio, la Universidad de California cubrirá el tratamiento médico necesario. Los costos del tratamiento pueden ser facturados a usted o su asegurador al igual que cualquier otro costo médico, o cubierto por la Universidad de California, dependiendo de una serie de factores. La Universidad normalmente no cubrirá ninguna otra forma de compensación por lesiones. Para obtener más información sobre esto, puede llamar a la oficina de la Junta de Revisión Institucional al 415-476-1814

Su firma a continuación indica que usted:

• Ha leído la información en este documento;

- Ha tenido la oportunidad de hacer cualquier pregunta que pueda tener sobre el estudio;
- Ha aceptado estar en el estudio y que su hijo esté en el estudio;
- Le han dicho que puede cambiar de opinión y retirar su consentimiento para participar en cualquier momento;
- Se le ha entregado una copia de la Carta de Derechos del Experimento Sindical para conservar y ha enviado por correo electrónico una copia de este formulario de consentimiento o una copia impresa;
- Le han dicho que al firmar el documento de consentimiento no renuncia a ninguno de sus derechos legales;
- Permite que el personal de investigación obtenga información de asistencia dental del software de mantenimiento de registros de Early Head Start; y,
- Permite que el personal de investigación obtenga datos de cepillado recogidos por la aplicación Sonicare y el cepillo de dientes de Philips Oral Healthcare. Estos datos incluyen: el momento en que comenzó el cepillado, la duración del cepillado, el cepillado conectado a la aplicación, el cepillado no conectado a la aplicación y la duración de la sesión de la aplicación.

Por favor también indique si desea que las imágenes orales (dentro de la boca del niño) de su hijo se usen para otros fines científicos después del final de este estudio.

| □ Acepto permitir que las imágenes orales de mi hijo se usen de forma anónima (no |
|---|
| vinculada) para otros estudios de investigación futuros. |
| □ No deseo que las imágenes orales de mi hijo se usen para otros estudios de |

investigación futuros.

También le pedimos que nos informe si no desea ser contactado en el futuro para su posible participación en otros programas de investigación.

- □ Acepto que me contacten para otros estudios de investigación futuros.
- □ No deseo ser contactado para otros estudios de investigación futuros.

| I INMA DEL PADRE O GUARDIAN LEGAL | FIRMA DEL PADRE O GUARDIAN LEG <i>i</i> | ۱L |
|---|---|---|
|---|---|---|

consentimiento y el permiso de los padres

| Nombre del niño | |
|---|---|
| Nombre del padre o guardián legal | <u> </u> |
| Firma del padre o guardián legal | Fecha |
| FIRMA DE LA PERSONA OBTENIENDO EL<br>PADRES | CONSENTIMIENTO Y EL PERMISO |
| Nombre de la persona obteniendo consentimiento y permiso del padre | Número de contacto |
| Firma de la persona que obtiene el | |

**DE LOS**